CLINICAL TRIAL: NCT06613412
Title: Feasibility and Safety of Remote Robotic Bronchoscopy System in Diagnosis of Peripheral Pulmonary Lesions: a Multicenter, Randomized Controlled, Proof-of Concept Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Li Shiyue, professor, Guangzhou Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: ES-2024-063-01
Record Dates: First submitted 2024-07-06; First posted 2024-09-26 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-07

CONDITIONS: Pulmonary Nodule
Keywords: peripheral pulmonary lesions; remote bronchoscopy; robotic bronchoscopy system

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (2):
- 5G group (Experimental): Biopsies of patients with pulmonary peripheral lesions (PPL) were performed using a remotely operated robotic bronchoscopy system supported by a 5G network.
  Interventions: Diagnostic Test: Remote Robotic Bronchoscopy system
- local group (No Intervention): In the absence of 5G network support, a local robotic bronchoscopy system is utilized to perform biopsies on patients with pulmonary peripheral lesions (PPL).

INTERVENTIONS:
Diagnostic Test: Remote Robotic Bronchoscopy system — Utilization of a remote robotic bronchoscopy system for the biopsy of patients with pulmonary peripheral lesions
  Arms: 5G group

SUMMARY:
Robotic bronchoscopy represents the latest localization technology for peripheral pulmonary nodules, enabling precise and stable manipulation, thereby enhancing the diagnostic yield of peripheral lung pathologies. Its safety and feasibility have been internationally validated, with indications that it can significantly improve the overall diagnostic rate of biopsies for peripheral lung lesions. Nonetheless, the disparity in interventional auxiliary equipment and the level of technical operation is the primary cause for the significant variation in diagnostic rates of peripheral lung lesions across different regions, particularly in remote or underdeveloped areas. The advancement of 5G network technology has propelled the development of telemedicine, enabling remote diagnostics, surgeries, and real-time multi-party collaboration, which is expected to elevate the medical standards in remote areas, improve the diagnostic rate of peripheral lung lesions, and achieve homogenization of medical services. In summary, the integration of 5G with bronchoscopy is anticipated to bring breakthroughs in the diagnosis and treatment of peripheral lung pathologies.

Research Objective:

The primary objective of this clinical trial is to evaluate the safety and efficacy of the remote application of bronchoscopy systems and catheters for the localization and sampling of peripheral pulmonary nodules, under the premise of ensuring the safety of the subjects and the scientific integrity of the clinical trial, with the aid of 5G network.

Research Method:

The study is a prospective, multicenter, single-arm clinical trial with a target value design, intending to include 10 cases of individuals with peripheral pulmonary nodules who are willing to undergo intra-airway examination and sampling operations using remote bronchial navigation localization devices assisted by the 5G communication network. The safety and efficacy of the bronchial navigation localization devices and catheters for the localization and sampling of peripheral pulmonary nodules, developed by Changzhou Langhe Medical Devices Co., Ltd. (hereinafter referred to as "Langhe Medical"), will be assessed.

Analysis:

Statistical data analysis will be performed using SAS software version 9.4 or higher.

DETAILED DESCRIPTION:
Study design

This study is a prospective, multicenter, single-group target value clinical trial, intending to include 10 cases of peripheral pulmonary nodules who are willing to accept airway examination and sampling operations assisted by a remote bronchoscopy system under the 5G communication network. The safety and efficacy of the bronchial navigation and localization equipment and catheter developed by Changzhou Langhe Medical Device Co., Ltd. (hereinafter referred to as 'Langhe Medical') for peripheral pulmonary nodule localization and sampling are evaluated.

The detailed operation of using the bronchial navigation and localization equipment and catheter for peripheral pulmonary nodule localization and sampling is as follows:

1. Conduct a network test before the experiment: Both test sites connect in advance to ensure that the network signal at the operation site meets the requirements.
2. Perform a chest CT examination on the patient, import the CT data into the system, mark the location of the target lesion, and plan the route;
3. Fasting for 6 hours before surgery and hydrating for 2 hours;
4. During the surgery, the patient is asked to lie flat, with the neck slightly hyperextended. Under general anesthesia, the glottis is exposed using a laryngoscope, and a tracheal intubation and ventilator-assisted ventilation are placed under direct vision. The main controller operator, assisted by the 5G network, remotely controls the co-controller's mechanical arm to make the bronchial navigation and localization equipment and catheter (hereinafter referred to as 'the catheter') pass through the tracheal intubation to the carina for navigation registration. After the registration is completed, under the continuous view of the catheter and real-time positioning guidance, precise control is achieved within the airway, and the planned route is followed through various bronchi, image collection is performed at each pulmonary segment opening, and the target lesion location is reached according to real-time navigation data;
5. When the lesion is visible under the field of view of the catheter's front-end camera, or when the co-controller operator confirms the arrival at the lesion through radial ultrasound via the catheter's working channel, after the researchers from both sites determine that the actual distance is sufficient to complete the biopsy sampling, the co-controller operator will send biopsy forceps, cell brushes, and other instruments through the catheter's working channel to complete the sampling by clamping and brushing;
6. Each subject collects 5-8 tissue specimens, which are processed for liquid-based cytology, smears, and pathology, and all specimens are sent for immediate pathological examination;
7. Postoperative follow-up to observe the occurrence of adverse events. The operation process must strictly follow the relevant operation specifications and be carried out according to the product instructions of the corresponding equipment. Accurate localization of the target pulmonary nodule, close observation of vital signs, presence of postoperative complications, and adverse events related to the test equipment should be maintained. Adverse events should be observed before discharge/discharge or within 3 days after the operation, and if respiratory distress symptoms occur, chest X-rays or other examinations should be conducted for confirmation.

ELIGIBILITY:
Inclusion Criteria:

Patients are eligible for inclusion if they meet all of the following criteria:

Age ≥18 years and ≤75 years, with no gender restrictions; Presence of a peripheral lung lesion on chest CT [Peripheral lung is defined as a nodule located in the fourth-order or higher airway (with the carina defined as order 0, the left and right main bronchi defined as order 1, lobar bronchi as order 2, segmental bronchi as order 3, and subsegmental bronchi as order 4)] in patients who require biopsy [2. The population requiring biopsy refers to individuals identified with an occupational lung lesion/nodule (including solid nodules, part-solid nodules, and ground-glass nodules) during clinical trial screening or with risk factors, and who, after comprehensive assessment by a clinician of the patient's clinical information, imaging, tumor markers, and functional imaging, are highly suspected of having cancerous nodules. Bronchoscopy biopsy is planned to further clarify the diagnosis and to guide staging treatment based on pathological results.]; Patients voluntarily agree to undergo bronchoscopy and meet the requirements for the procedure; Patients are capable of understanding the purpose of the trial, demonstrate good compliance with the examinations and follow-up, voluntarily participate in the clinical trial, and sign an informed consent form.

-

Exclusion Criteria:

Patients who meet any of the following criteria will be excluded from this study:

1.Presence of contraindications for bronchoscopy, including: active massive hemoptysis; recent myocardial infarction or unstable angina; severe cardiac or pulmonary dysfunction; severe hypertension and arrhythmias; uncorrectable bleeding tendencies or severe coagulation disorders (such as platelet count <60×10^9/L), uremia; severe pulmonary artery hypertension; severe superior vena cava syndrome; intracranial hypertension; acute cerebrovascular events; aortic dissection or aneurysm; multiple bullae; extreme systemic exhaustion; 2.Female patients who are breastfeeding, pregnant, or planning pregnancy; 3.Patients with electromagnetic active implantable medical devices; 4.Subjects allergic to anesthetics; or with a history of multiple severe allergies, hereditary allergy history; 5.Those who have participated in or are currently participating in drug clinical trials within 3 months before screening, or have participated in other medical device clinical trials within 30 days; 6.Any other conditions deemed unsuitable for participation in this clinical trial by the investigator.

-

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-09-15 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-02-15 (Estimated)

PRIMARY OUTCOMES:
equipment failure rate | During the bronchoscopy
  The equipment failure rate is calculated as (number of instances of equipment failure / total number of uses) x 100%. Equipment failures are defined as follows: 1. Network delays ≥ 200ms that persist for more than 3 seconds; 2. Any equipment malfunction that results in the cessation of surgery.

SECONDARY OUTCOMES:
Average Latency | During the operation
  Refers to the network data transmission delay, recording the continuous latency data from the start of registration to the end of sampling, and documenting the average, peak, and minimum values.
Bandwidth | During the operation
  Refers to the network transmission rate, recording the network bandwidth from the start of registration to the end of sampling at both control ends, documenting the maximum upload and download bandwidth.
Network Incidents and Recovery Time | During the operation
  Records the specific incidents and quantities of network interruptions and individual stutters >10 seconds during a single operation.
Sampling yield | 7 days after bronchoscopy
  Sampling yield = (Total number of cases with non-normal lung tissue obtained by biopsy sampling / Total number of cases undergoing biopsy sampling) × 100%. Note: Definitive sampling includes biopsy pathological results indicating cells/tissues as malignant, benign lesions (such as fungi, tuberculosis, or sarcoidosis, etc.), and non-normal lung tissue that cannot be confirmed.
Incidence of Adverse Events | 7 days after operation
  Incidence of Adverse Events= (Number of cases with adverse events / Total number of sampled cases) × 100%
  Definitive adverse events includes: (1) any type of pneumothorax, irrespective of the necessity for tube thoracostomy, (2) bleeding during bronchoscopy requiring intervention, and (3) other adverse events such as fever, pain, and cough.

OTHER OUTCOMES:
Diagnostic yield | 7 days after bronchoscopy
  Diagnostic yield is defined as the proportion of cases diagnosed with bronchoscopy pathology divided by all cases sampled using a specific technology. The bronchoscopy pathology diagnosis only included malignant and specific benign lesions. A lesion was considered malignant if tumor cells were found in histological and/or cytological specimens. Specific benign findings included granuloma, organizing pneumonia, purulence or robust neutrophilic inflammation, and other less common specific benign findings such as those suggesting hamartoma or amyloidoma.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Skouras VS, Gkiozos I, Charpidou AG, Syrigos KN. Robotic Bronchoscopy in Lung Cancer Diagnosis. Cancers (Basel). 2024 Mar 17;16(6):1179. doi: 10.3390/cancers16061179. PMID 38539514
- [Background] Huang J, Lin J, Chen C, Liang W, Chen Y, Li H, Zhong C, Li S. 5G-Based Remote Virtual Bronchoscopic Navigation-Guided Transbronchial Lung Biopsy for Diagnosis of Lung Cancer: Description of 2 Cases. Respiration. 2023;102(10):912-917. doi: 10.1159/000533867. Epub 2023 Oct 6. PMID 37806300